CLINICAL TRIAL: NCT06854250
Title: Androgen Deprivation Therapy Combined With Novel Androgen Receptor Inhibitors, Prostate Cryoablation, and Cyclophosphamide in the Treatment of Newly Diagnosed, Metastatic Prostate Cancer: A Single-Center, Single-Arm, Prospective Clinical Study
Brief Title: Prostate Cryoablation Combined With Metronomic Cyclophosphamide for Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Associate Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-295; SL-B2024-623-02 (Other: Sun Yst-sen University Cancer Center)
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic prostate cancer; Novel androgen receptor inhibitors; Prostate cryoablation; Cyclophosphamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cryoablation and cyclophosphamide (Experimental): Metastatic prostate cancer patients receive prostate cryoablation and metronomic cyclophosphamide in addition to androgen deprivation therapy and novel androgen receptor inhibitors.
  Interventions: Procedure: Prostate cryoablation; Drug: Cyclophosphamide (CTX)

INTERVENTIONS:
Procedure: Prostate cryoablation — Enrolled patients will receive prostate cryoablation within 6 months of starting androgen deprivation therapy.
Drug: Cyclophosphamide (CTX) — Enrolled patients will receive cyclophosphamide (50mg daily) one day after prostate cryoablation and continue for a total of six months.

SUMMARY:
The goal of this clinical trial is to explore whether androgen deprivation therapy combined with novel androgen receptor inhibitors, prostate cryoablation, and metronomic cyclophosphamide is superior to the current treatment regimen of androgen deprivation therapy plus novel androgen receptor inhibitors for patients with metastatic prostate cancer. It will also learn about the safety of prostate cryoablation, and metronomic cyclophosphamide for patients with metastatic prostate cancer. The main questions it aims to answer are:

Does prostate cryoablation, and metronomic cyclophosphamide delay the progression of metastatic prostate cancer? Does prostate cryoablation, and metronomic cyclophosphamide reduce symptomatic local events of metastatic prostate cancer?

Researchers will explore if androgen deprivation therapy combined with novel androgen receptor inhibitors, prostate cryoablation, and metronomic cyclophosphamide works to treat metastatic prostate cancer.

Participants will:

Receive treatment of androgen deprivation therapy and novel androgen receptor inhibitors until progression.

Receive prostate cryoablation surgery and take cyclophosphamide. Visit the clinic every 1-3 months for checkups and tests. Keep a diary of their symptoms.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of combining prostate cryoablation and cyclophosphamide with androgen deprivation therapy plus novel androgen receptor inhibitors (apalutamide, rezvilutamide, or darolutamide) in patients with newly diagnosed, metastatic prostate cancer. By comparing with previous studies, it seeks to explore whether prostate cryoablation and cyclophosphamide treatment can confer survival benefits and reduce symptomatic local urinary events in these patients.

Patients with newly diagnosed, metastatic prostate cancer who meet the inclusion criteria after evaluation will receive treatment with androgen deprivation therapy plus a novel androgen receptor inhibitor (apalutamide, rezvilutamide, or darolutamide) in combination with prostate cryoablation and cyclophosphamide. Enrolled patients should start the novel androgen receptor inhibitor (apalutamide, rezvilutamide, or darolutamide) within 3 months of initiating androgen deprivation therapy and undergo prostate cryoablation within 6 months of starting androgen deprivation therapy. Cyclophosphamide treatment will begin one day after prostate cryoablation and continue for a total of six months.

The primary endpoint of the study is PSA progression-free survival. Secondary endpoints include: 1) radiographic progression-free survival, 2) time to progression to metastatic castration-resistant prostate cancer, 3) overall survival, 4) PSA nadir, 5) incidence of symptomatic local events, and 6) safety.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 80 years old;
* Histopathological confirmation of prostatic acinar adenocarcinoma;
* Diagnosed with metastatic prostate cancer at initial diagnosis according to the AJCC 8th edition staging criteria;
* No progression at the time of initiating of prostate cryoablation;
* ECOG score of 0-1;
* Can tolerate general anesthesia and prostate cryoablation surgery;
* No significant abnormalities .
* Able to understand this study and sign the informed consent form.

Exclusion Criteria:

* Serious illness not suitable to receive the treatment regimen;
* Other malignant tumors (within 5 years), except for non-melanoma skin cancer;
* Receipt of treatments other than treatment regimen of this study;
* Prostate cancer invading the rectum;
* with prostate volumegreater than 55ml after 6 months of androgen deprivation therapy .

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
PSA progression-free survival | From date of initiation of androgen deprivation therapy until the date of PSA progression or date of death from any cause, whichever came first, assessed up to 5 years
  Defined as the time from the initiation of androgen deprivation therapy to the occurrence of PSA progression or death.

SECONDARY OUTCOMES:
Radiographic progression-free survival | From date of initiation of androgen deprivation therapy until the date of radiographic progression or date of death from any cause, whichever came first, assessed up to 5 years
  Defined as the time from the initiation of androgen deprivation therapy to the occurrence of radiographic progression of death.
mCRPC-free survival | From date of initiation of androgen deprivation therapy until the date of progression to metastatic castration-resistant prostate cancer or date of death from any cause, whichever came first, assessed up to 5 years
  Defined as the time from the initiation of androgen deprivation therapy to progression to metastatic castration-resistant prostate cancer (mCRPC) or death.
Overall survival | From date of initiation of androgen deprivation therapy until the date of death from any cause, assessed up to 5 years
  Defined as the time from the initiation of androgen deprivation therapy to death from any cause.
Incidence of symptomatic local events | Through study completion, an average of 3 year
  Symptomatic local events are defined as any of the following conditions: urinary tract infection, indwelling catheterization, acute kidney injury, transurethral resection of the prostate, urinary obstruction, indwelling ureteral stent placement, nephrostomy, colostomy, or surgery for intestinal obstruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Si T, Guo Z, Hao X. Combined cryoablation and GM-CSF treatment for metastatic hormone refractory prostate cancer. J Immunother. 2009 Jan;32(1):86-91. doi: 10.1097/CJI.0b013e31818df785. PMID 19307997
- [Background] Donnelly BJ, Saliken JC, Brasher PM, Ernst SD, Rewcastle JC, Lau H, Robinson J, Trpkov K. A randomized trial of external beam radiotherapy versus cryoablation in patients with localized prostate cancer. Cancer. 2010 Jan 15;116(2):323-30. doi: 10.1002/cncr.24779. PMID 19937954
- [Background] Shah TT, Peters M, Eldred-Evans D, Miah S, Yap T, Faure-Walker NA, Hosking-Jervis F, Thomas B, Dudderidge T, Hindley RG, McCracken S, Greene D, Nigam R, Valerio M, Minhas S, Winkler M, Arya M, Ahmed HU. Early-Medium-Term Outcomes of Primary Focal Cryotherapy to Treat Nonmetastatic Clinically Significant Prostate Cancer from a Prospective Multicentre Registry. Eur Urol. 2019 Jul;76(1):98-105. doi: 10.1016/j.eururo.2018.12.030. Epub 2019 Jan 9. PMID 30638633
- [Background] Tsuboi I, Matsukawa A, Kardoust Parizi M, Klemm J, Mancon S, Chiujdea S, Fazekas T, Miszczyk M, Laukhtina E, Kawada T, Katayama S, Iwata T, Bekku K, Karakiewicz P, Wada K, Roupret M, Araki M, Shariat SF. A Systematic Review and Meta-analysis of the Impact of Local Therapies on Local Event Suppression in Metastatic Hormone-sensitive Prostate Cancer. Eur Urol Oncol. 2024 Dec;7(6):1185-1194. doi: 10.1016/j.euo.2024.03.007. Epub 2024 Apr 4. PMID 38575408
- [Background] Li Y, Wang N, Zhao D, Wang J, Jiang L, Wang Y, Chen D, Wu Z, Zhou F, Yang Z. Cytoreductive prostate cryoablation and metronomic cyclophosphamide for metastatic hormone-sensitive prostate cancer. Future Oncol. 2022 Jun;18(19):2373-2380. doi: 10.2217/fon-2021-1424. Epub 2022 Apr 20. PMID 35440168
- [Background] Wang N, Ye Y, Deng M, Zhao D, Jiang L, Chen D, Wu Z, Wang Y, Li Z, Yang Z, Li J, Zhou F, Li Y. Prostate cryoablation combined with androgen deprivation therapy for newly diagnosed metastatic prostate cancer: a propensity score-based study. Prostate Cancer Prostatic Dis. 2021 Sep;24(3):837-844. doi: 10.1038/s41391-021-00335-2. Epub 2021 Mar 4. PMID 33664457